CLINICAL TRIAL: NCT02504866
Title: Effect of Exercise Training on Physical, Cognitive and Behavioral Function in Patients With Traumatic Brain Injury
Brief Title: Effect of Exercise Training on Physical, Cognitive, and Behavioral Function in People With TBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated early due to the COVID-19 pandemic.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 150164; 15-CC-0164
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-02

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: Aerobic Exercise Training; Balance; TBI; Rapid-Resistive Exercise
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Intervention (AET) (Experimental): Participant with traumatic brain injury performed aerobic exercise on an elliptical trainer at a vigorous intensity for 30 minutes three times a week for 12 weeks
  Interventions: Other: Vigorous exercise
- Rapid-Resistive Exercise Intervention (RET) (Experimental): Participant with traumatic brain injury performed rapid reciprocal exercise on an elliptical trainer at light to moderate intensity for 30 minutes three times a week for 12 weeks
  Interventions: Other: Light to moderate exercise
- Waitlist Control (CON) (No Intervention): Participant with traumatic brain injury were waitlisted and did not perform any exercise intervention in the first 12 weeks. They were randomized to either AET or RET after the initial 12 weeks

INTERVENTIONS:
Other: Vigorous exercise — Exercise training of vigorous intensity
  Arms: Aerobic Exercise Intervention (AET)
Other: Light to moderate exercise — Exercise training of light to moderate intensity
  Arms: Rapid-Resistive Exercise Intervention (RET)

SUMMARY:
Background:

- Traumatic brain injury (TBI) often causes problems with moving and balance, and thinking and emotions. Exercise can improve these things in people with other brain damage. Researchers want to look at the effect of exercise on these things in people with TBI.

Objectives:

- To study how head injuries affect the brain. To study if exercise can help some symptoms in people with TBI. These include problems thinking, balancing, and moving, and depression or anxiety.

Eligibility:

* People age between 18 and 79
* Had a non-penetrating TBI at least 12 months ago
* Are physically inactive, but can stand and walk without help

Design:

* Participants will be screened with medical history, physical exam, and blood and urine tests. They may have a balance test.
* Participants will be assigned to a high-intensity or a lower-intensity exercise program.
* The study is 6 months long. There will be 3 months with exercise on an elliptical machine and 3 months without exercise.
* Participants will exercise for 30 minutes on an elliptical machine, 3 days per week for 3 months.
* Participants will also have 3 outpatient testing visits lasting approximately 8 hours, once every 3 months. This visit will include:
* Blood tests
* Tests for memory, attention, and thinking
* Tests of walking and balance
* Questionnaires
* An MRI: they will lie in a machine that takes pictures of their brain, while breathing regular air and air with more carbon dioxide
* Test of physical fitness

DETAILED DESCRIPTION:
Objective

The broad objective of this study is to examine the effects of moderate and more intense aerobic exercise as an intervention on cognitive performance, physical functioning and health-related quality of life in patients with chronic (more than 12 months post-injury) traumatic brain injury (TBI). Importantly, structural and biological brain changes will be measured to examine whether functional outcomes are related to exercise-induced adaptations. It is hypothesized that in the chronic phase of persons with TBI, there will be improved: 1) cognitive function, 2) physical fitness and fatigue severity, 3) motor performance and balance, and 4) mood and depressive symptoms, in those that performed the exercise intervention compared to a control group. It is also hypothesized that these functional improvements will be related to exercise intensity, improved cortical connectivity, dopamine transmission gene scores, and blood biomarkers related to neuro and angio-genesis.

Study Population

80 ambulatory adults with non-penetrating TBI will be enrolled. We will also enroll up to 20 healthy volunteers as a comparison group for some of the outcome measures. Subjects will be recruited from NIH, affiliated hospitals/clinics and the community

Design

Healthy volunteers will have a limited assessment that includes brain imaging, blood draw for genetic testing, and a subset of the cognitive and behavioral testing at a single time-point. All subjects with TBI will perform baseline assessments including cognitive and behavioral performance, brain imaging, fitness, motor and balance testing, and selected blood and genetic testing. Thereafter, subjects with TBI will be randomized to either a waitlist control, or one of two exercise conditions: 1) 30 minutes at a fast pace, moderate-intensity (rapid-resistive exercise; RET); 2) 30 minutes at higher-intensity (aerobic exercise; AET). Both exercise groups will perform the exercise on an elliptical trainer 3 times a week, for a session duration of 45 minutes including warm-up and cool-down. The RET group will focus on rapid reciprocal motion with minimal resistance, while the AET group will exercise at an elevated intensity known to produce an aerobic effect. After 12 weeks, all groups will repeat the baseline assessments (3 month follow-up). Following this assessment, the waitlist control group will be randomized to either RET or AET and the exercise groups will cease formal supervised exercise sessions. A third assessment visit will be performed after an additional 12 weeks (6 month follow-up).

Outcome Measures

Cognitive performance will be tested and interpreted compared to norms. Performance on motor and balance tasks will be assessed with the Smart Balance Measurement System and the GAITRite System. Physical fitness will be determined by peak oxygen consumption and aerobic threshold as measured by pulmonary gas exchange during an exercise tolerance test on the treadmill. Structural brain volumes will be determined by magnetic resonance imaging (MRI) and cortical connectivity will be quantified using resting state functional MRI and Diffusion Tensor Imaging (DTI) to evaluate integrity of and changes in white matter tracts in response to exercise and compared to healthy volunteers. Blood will be collected to quantify the presence of biomarkers (such as VEGF, BDNF and IGF-1) and dopamine transmission. Other self-reported measures of quality of life, fatigue severity, depression and sleep quality would also be collected, and compared to healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for those with TBI:

1. Ages 18 to 79 inclusive
2. Diagnosis of non-penetrating TBI
3. Injury occurred at least 12 months prior to enrollment
4. Physically inactive as identified by a physician
5. Able to stand and walk independently and safely without any assistance
6. Able to follow the study protocol
7. Fluent in English and able to provide informed consent

Inclusion criteria for healthy volunteers:

1. Ages 18 to 79 inclusive
2. Physically inactive as identified by a physician
3. Fluent in English

EXCLUSION CRITERIA:

Exclusion criteria for those with TBI:

1. History of exercise intolerance
2. History of heart disease
3. History of pulmonary disease, other than controlled, non-exercise-induced asthma
4. History of uncontrolled diabetes
5. Uncontrolled hypertension, defined as a resting blood pressure > 140/90 mmHg
6. On medications that would influence aerobic capacity or treadmill performance such as beta blockers or antiretroviral therapy
7. Active substance abuse including ETOH
8. Presence of an injury to any extremity, or other medical condition that would affect motor function or the ability to perform the assessment or the exercise program, specifically balance problems due to vestibulopathy
9. Unable to refrain from smoking at least 4 hours prior to exercise testing sessions
10. Medical or psychological instability such that the subject could not reasonably be expected to fulfill the study requirements
11. Pregnancy
12. BMI >40 kg/M(2) due to the limits of the treadmill, elliptical machine and MRI scanner
13. Planning to make a change in medication or therapy during the enrollment period with the goal of improving mood, cognitive function or motor function
14. Have any of the following contraindications to having an MRI scan:

    1. A ventriculo-peritoneal shunt
    2. Have claustrophobia and not comfortable in small enclosed spaces
    3. Have metal that would make an MRI scan unsafe such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion devise, cochlear or ear implant, transdermal medication patch (nitroglycerine), any metallic implants or objects, body piercing that cannot be removed, bone or joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal embedded (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near your eyes).
    4. Excessive startle reaction to or fear of loud noises

Exclusion criteria for healthy volunteers:

1. History or presence of cardiopulmonary or respiratory disease
2. History or presence of other disease of the neurologic, metabolic, or renal systems
3. Active substance abuse including ETOH
4. Pregnancy
5. BMI >40 kg/m2
6. Medical or psychological instability such that the subject could not reasonably be expected to fulfill the study requirements
7. Have any contraindications to having an MRI scan

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and samples will be stored in the Center for Neuroscience and Regenerative Medicine (CNRM) data and biospecimen repositories, respectively. Data uploaded to the CNRM repository will be made available to other CNRM researchers upon request.
Supporting Information: Study Protocol, ICF
Access Criteria: The Data Quality, Access, and Publication Committee will be responsible for procedures for Center for Neuroscience and Regenerative Medicine (CNRM) investigators to provide the necessary information for review of investigator qualifications and data usage. CNRM investigators requesting data must submit documentation of Institutional Review Board (IRB) approval of the research project with consideration of approvals across multiple sites if applicable. Only de-identified data can be requested. Use of the data is limited to the project that was proposed and approved. The data may not be reused for other projects or analyses, or redistributed to other investigators, repositories or databases, without written approval from the CNRM Data Quality, Access, and Publication Committee and the CNRM Informatics Core. At the completion of the analysis, the data and results must be entered into the CNRM repository.

REFERENCES:
- [Background] Chin LM, Keyser RE, Dsurney J, Chan L. Improved cognitive performance following aerobic exercise training in people with traumatic brain injury. Arch Phys Med Rehabil. 2015 Apr;96(4):754-9. doi: 10.1016/j.apmr.2014.11.009. Epub 2014 Nov 26. PMID 25433219
- [Background] Chin LM, Chan L, Woolstenhulme JG, Christensen EJ, Shenouda CN, Keyser RE. Improved Cardiorespiratory Fitness With Aerobic Exercise Training in Individuals With Traumatic Brain Injury. J Head Trauma Rehabil. 2015 Nov-Dec;30(6):382-90. doi: 10.1097/HTR.0000000000000062. PMID 24901330
- [Background] Damiano DL, Zampieri C, Ge J, Acevedo A, Dsurney J. Effects of a rapid-resisted elliptical training program on motor, cognitive and neurobehavioral functioning in adults with chronic traumatic brain injury. Exp Brain Res. 2016 Aug;234(8):2245-52. doi: 10.1007/s00221-016-4630-8. Epub 2016 Mar 30. PMID 27025506
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-CC-0164.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 20 subjects consented, four subjects withdrew prior to being randomized, five subjects were screen failures.
  Three of the four subjects from the Waitlist Control arm (CON) were further randomized to either AET or RET
Groups:
- Waitlist Control (CON): Participant with traumatic brain injury were waitlisted and did not perform any exercise intervention in the first 12 weeks. They were randomized to either Aerobic Exercise Intervention (AET) or Rapid-Resistive Exercise Intervention (RET) after the initial 12 weeks.
Period: 3-Month Follow up
Arm/Group | Aerobic Exercise Intervention (AET) | Rapid-Resistive Exercise Intervention (RET) | Waitlist Control (CON)
Started | 4 | 3 | 4
Completed | 4 | 3 | 4
Not Completed | 0 | 0 | 0
Period: 6-Month Follow up (CON Group Only)
Arm/Group | Aerobic Exercise Intervention (AET) | Rapid-Resistive Exercise Intervention (RET) | Waitlist Control (CON)
Started | 1 (First period was CON arm) | 2 (First period was CON arm) | 0
Completed | 0 | 2 | 0
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise Intervention (AET) | Rapid-Resistive Exercise Intervention (RET) | Waitlist Control (CON) | Total
Number analyzed (Participants) | 4 | 3 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 10
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 4
  Male | 1 | 2 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 2 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 2 | 2 | 7
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function as Measured by Trail Making Test Part B (TMT-B)
Description: Trail Making Test (TMT) is a neuropsychological assessment of visual conceptual and visual motor tracking (involves motor speed and attention functions). Trail Making Test Part B (TMT-B) is associated with executive functioning and involves drawing a line connecting alternating numbers and letters in sequence (i.e., 1-A-2-B and so on). The time to complete the test is recorded. The time taken to complete the test was converted into standardized T-scores, representing a mean of 50 and a standard deviation of 10. Higher T-scores mean less cognitive deficits. The change in cognitive function was reported as the change in TMT-B T-scores across the 12 weeks (post minus pre intervention).
Time Frame: Before (pre) and after (post) 12 weeks intervention
Population: The analyses included only those subjects who completed TMT-B at baseline and 3-month follow-up time points.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Aerobic Exercise Intervention (AET) | Rapid-Resistive Exercise Intervention (RET) | Waitlist Control (CON)
Number analyzed (Participants) | 4 | 3 | 4
T-score | 4.5 (3.7) | -6.33 (29.02) | -6.75 (17.17)

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Waitlist Control (CON): Participant with traumatic brain injury were waitlisted and did not perform any exercise intervention in the first 12 weeks.
Arm/Group | Aerobic Exercise Intervention (AET) | Rapid-Resistive Exercise Intervention (RET) | Waitlist Control (CON)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/5 | 2/5 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Intervention (AET) (N=5) | Rapid-Resistive Exercise Intervention (RET) (N=5) | Waitlist Control (CON) (N=4)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise Intervention (AET) (N=5) | Rapid-Resistive Exercise Intervention (RET) (N=5) | Waitlist Control (CON) (N=4)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
hypoglycaemia (Endocrine disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0
suicidal ideation (Psychiatric disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early due to the COVID-19 pandemic. Enrollment of subjects were suspended, then major equipment changes and infection control updates precluded continuation during the COVID-19 pandemic. No subjects were enrolled into the healthy volunteer arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT02504866/Prot_SAP_000.pdf